CLINICAL TRIAL: NCT01865656
Title: Skills and Drills Intervention for Improving Emergency Obstetric and Neonatal Care in Select First Referral Units in Northern Karnataka
Brief Title: A Skills and Drills Intervention for Emergency Obstetrics and Neonatal Care at First Referral Units of North Karnataka
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: St. John's Research Institute (Other); Maternal Health Task Force (Unknown); Bill and Melinda Gates Foundation (Other); Karnataka Health Promotion Trust (Other)
Responsible Party: Principal Investigator, Ana Langer, Director of the Women and Health Initiative, Harvard School of Public Health (HSPH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MHTF IR India; REF/2013/05/005058 (Registry Identifier: Clinical Trials Registry- India)
Record Dates: First submitted 2013-05-28; First posted 2013-05-31 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Obstetric and Perinatal Complications; Postpartum Hemorrhage; Preeclampsia/Eclampsia; Obstructed/Prolonged Labor; Sepsis; Birth Asphyxia
Keywords: provider skill and self-efficacy; Appropriate and timely referral for obstetric emergencies; Intervention feasibility and acceptability
MeSH Terms: conditions — Postpartum Hemorrhage; Pre-Eclampsia; Eclampsia; Sepsis; Asphyxia Neonatorum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 4 intervention first referral units (Other): A Quasi-experimental intervention/control trial will be implemented to assess the impact of the following interventions on the outcome measures in a cluster of 4 intervention sites relative to a matched cluster of 4 control sites:
  Refresher/simulation training to improve provider skills/knowledge Implementation of Emergency Obstetric Drills Revised Case sheets(for data collection and therefore part of both control and intervention sites), Mentoring and Supportive supervision, and Referral Strengthening
  Interventions: Other: Skills training; Other: Emergency obstetric drills; Other: Revised Case Sheets; Other: Supportive supervision; Other: Referral strengthening
- Control Arm (No Intervention)

INTERVENTIONS:
Other: Skills training — Refresher training on Basic Emergency Obstetric and Newborn care
  Arms: 4 intervention first referral units
Other: Emergency obstetric drills — Emergency obstetric drills to practice timely and appropriate management of postpartum hemorrhage and preeclampsia/eclampsia
  Arms: 4 intervention first referral units
Other: Revised Case Sheets — Revised case sheets will be introduced to capture the timing and appropriate medical treatment of women in labor and newborns
  Arms: 4 intervention first referral units
Other: Supportive supervision — Quarterly supportive supervision visits each of the intervention first referral units.
  Arms: 4 intervention first referral units
Other: Referral strengthening — To support referral systems that ensure timely and appropriate treatment for obstetric emergencies
  Arms: 4 intervention first referral units

SUMMARY:
To evaluate the effectiveness of a First Referral Unit (FRU) Emergency Obstetric and Newborn Care (EmONC) skills and drills intervention, to estimate the appropriateness and effectiveness of referrals in intervention arm compared to control arm and to calculate the incremental cost and cost effectiveness of EmONC skills and drills intervention.

DETAILED DESCRIPTION:
The aim of this intervention is to improve the quality of care for institutional births with a special focus on improving the quality of Emergency Obstetric and Newborn Care (EmONC). This intervention will focus on improving the skills and practices of providers and through the improvement of referral networks, ensure timely and appropriate management of complications.

The specific objectives include:

1. Evaluate the effectiveness of an FRU-level Basic and EmONC Skills and Drills intervention combined with the existing primary health centre (PHC) based nurse mentoring intervention in improving appropriate diagnosis and management of obstetric and perinatal complications.
2. Assess the additional benefit of the EmONC Skills and drills intervention at FRUs in terms of improvement of obstetric and perinatal outcomes compared to the PHC-level intervention alone.
3. Estimate the appropriateness and effectiveness of referrals in intervention facilities compared to controls.
4. Calculate the incremental cost and cost-effectiveness of the EmONC skills and drills intervention

ELIGIBILITY:
Inclusion Criteria:

All women age who are referred or admitted directly to the first referral unit for a delivery or with a complication Staff working in the First Referral Units

Exclusion Criteria:

no specific exclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15018 (Actual)
Dates: Start 2013-07; Primary Completion 2014-10 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Appropriate management of direct obstetric and perinatal complications | Month 18 of the project
  Appropriate and timely management of postpartum hemorrhage (PPH), Preeclampsia, Obstructed or prolonged labor, Sepsis and birth asphyxia

SECONDARY OUTCOMES:
Feasibility of the intervention | Month 18 of the project
  We will evaluate barriers and facilitators of implementing these intervention packages, as well as costing them.
Acceptability of the intervention | Month 18 of the project
  Using in-depth interviews with providers, we will assess the acceptability of the interventions.
Self-efficacy of health care personnel to manage direct obstetric and neonatal complications | Month 18 of the project
  Providers will be assessed on self-efficacy pre and post intervention
Knowledge and skills competency of health care personnel on the management of obstetric and neonatal complications | Month 18 of the project
Case-fatality rates | Month 18 of the project
  Using data from obstetric and newborn case sheets we will assess case-fatality rates
Timeliness and appropriateness of referral | Month 18 of the project

CONTACTS AND LOCATIONS:
Overall Officials: Beena Verghese, PhD, Principal Investigator — St. John's Research Institute, Public Health Foundation of India; Prem Mony, MD, MSc, Principal Investigator — St. John's Research Institute, Bangalore; Krishnamurthy Jeyanna, MD, Principal Investigator — Karnataka Health Promotion Trust; Ana Langer, MD, Principal Investigator — Harvard School of Public Health (HSPH); Fernando Althabe, MD, Principal Investigator — Institute for Clinical Effectiveness and Health Policy